CLINICAL TRIAL: NCT05836246
Title: The Development of Artificial Intelligence (AI) Based High Performance Structural-functional and Quantitative Ultrasound Imaging Software Platform
Brief Title: The Development of Quantitative Ultrasound Imaging Software Platform
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-1910-570-301
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Chronic Liver Disease; Thyroid Disease; Benign Breast Disease; Malignant Breast Neoplasm; Acute Myocardial Infarction
MeSH Terms: conditions — Thyroid Diseases; Cystic Fibrosis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare the image differences between conventional ultrasound and artificial intelligence-based ultrasound software in conscious adults.

The main question it aims to answer is to evaluate the effectiveness by determining that the new image analysis method is considered valid if it helps to identify more than 30% of histological characteristics.

Participants will undergo the examination using the two methods mentioned earlier after signing the consent form.

ELIGIBILITY:
Inclusion Criteria:

* People with heart disease, thyroid disease, breast disease, and liver disease.

Exclusion Criteria:

* Someone who has received surgery on the target organ in question.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A person who visits Seoul National University Bundang Hospital for medical treatment or consultation.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative ultrasound information | 5 years
  Quantitative ultrasound images of heart, thyroid, and breast disease

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Cheng PM, Malhi HS. Transfer Learning with Convolutional Neural Networks for Classification of Abdominal Ultrasound Images. J Digit Imaging. 2017 Apr;30(2):234-243. doi: 10.1007/s10278-016-9929-2. PMID 27896451
- [Result] Chi J, Walia E, Babyn P, Wang J, Groot G, Eramian M. Thyroid Nodule Classification in Ultrasound Images by Fine-Tuning Deep Convolutional Neural Network. J Digit Imaging. 2017 Aug;30(4):477-486. doi: 10.1007/s10278-017-9997-y. PMID 28695342
- [Result] F. Milletari, N. Navab and S. -A. Ahmadi. V-Net: Fully Convolutional Neural Networks for Volumetric Medical Image Segmentation. 2016 Fourth International Conference on 3D Vision (3DV), Stanford, CA, USA. 2016; 565-571.
- [Result] Ma J, Wu F, Jiang T, Zhu J, Kong D. Cascade convolutional neural networks for automatic detection of thyroid nodules in ultrasound images. Med Phys. 2017 May;44(5):1678-1691. doi: 10.1002/mp.12134. Epub 2017 Apr 17. PMID 28186630
- [Result] Chen H, Zheng Y, Park JH, Heng PA, Zhou SK. (2016). Iterative Multi-domain Regularized Deep Learning for Anatomical Structure Detection and Segmentation from Ultrasound Images. Medical Image Computing and Computer-Assisted Intervention - MICCAI 2016. 2016; 9901.
- [Result] Lekadir K, Galimzianova A, Betriu A, Del Mar Vila M, Igual L, Rubin DL, Fernandez E, Radeva P, Napel S. A Convolutional Neural Network for Automatic Characterization of Plaque Composition in Carotid Ultrasound. IEEE J Biomed Health Inform. 2017 Jan;21(1):48-55. doi: 10.1109/JBHI.2016.2631401. Epub 2016 Nov 22. PMID 27893402